CLINICAL TRIAL: NCT02802384
Title: Investigation of Pathophysiology of Angiogenesis and Osteogenesis in Paget's Disease of Bone
Brief Title: Pathophysiology of Paget's Disease of Bone
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00077130
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Paget's Disease of Bone
Keywords: Paget's Disease of Bone; Healthy controls
MeSH Terms: conditions — Osteitis Deformans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human blood samples with be collected. One tube of blood will be utilized to measure specific serum chemokine concentrations. One tube will be utilized to extract DNA for potential future studies if permission is provided. The remainder of the blood sample will be utilized to count the number of stem cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: People with active Paget's Disease of Bone
- Controls: Age and sex matched people without history of Paget's Disease of Bone

SUMMARY:
Paget's disease of the bone is a skeletal disorder which results in increased and disorganized bone remodeling, leading to dense but fragile and expanding bones. The identified genetic causes of Paget's disease of bone only explain why bone is destroyed, but not why the bone formed in its place is abnormal.

Current treatment for people with Paget's disease of the bone is limited to patients with bone pain, thought to be related to high rate of bone turnover (breakdown and rebuilding of bone) and works by slowing down the rate of bone breakdown. The current treatment does not address the excess blood vessels and bone formed.

This research is being done to understand factors that may promote blood vessel and bone formation in Paget's disease of the bone.

DETAILED DESCRIPTION:
The genetic mutations found in Paget's disease currently only account for about 15% of cases and are limited to genes that affect osteoclast differentiation and function. These mutations alone are insufficient to explain the full phenotype, particularly hypervascularity and increased bone formation. Through a series of basic science studies, the investigators have recently found that preosteoclasts secrete chemokines to promote migration of various stem cells, which then differentiate into osteoblasts and endothelial cells to support osteogenesis and angiogenesis, respectively.

The investigators will perform a cross sectional study of patients with active Paget's disease of bone compared to similar people without Paget's disease of bone. The goal is to enroll 10 patients with Paget's disease of the bone (cases) and 10 healthy, age- and sex-matched people (controls) whom meet similar exclusion criteria. Participants who consent to the study will undergo a brief history and physical exam, allow review of medical records relevant to their disease, and have one blood (5 tablespoons) sample drawn.

The investigators hypothesize that specific chemokine concentrations are increased in people with Paget's disease of the bone compared to controls. The investigators also hypothesize that these levels correlate with severity of disease. Therefore, the investigators primary objective is to determine if serum chemokine levels are increased in patients with Paget's disease of the bone. The secondary objective is to evaluate if the serum chemokine concentrations correlate with various markers of disease activity. Findings could aid in the clinical monitoring of patients with Paget's disease of the bone and could provide an additional therapeutic target to improve treatment of this painful disease.

ELIGIBILITY:
Inclusion Criteria for Cases:

* Men and women between the ages of 18-99 years who have evidence of active Paget's disease of bone as clinically and/or radiographically defined by:

  * Increased serum alkaline phosphatase or increased serum collagen type 1 c-telopeptide (CTX) or increase in urinary pyridinoline at diagnosis
  * AND history of at least one of the following signs/symptoms: Pagetoid lesions(s) on x-ray/CT/MRI, increased uptake of radioactive substance by bone scan, bone pain, fracture, hearing loss, headache, hypercalcemia, or bony deformity.

Inclusion criteria for controls:

* Men and women between the ages of 18-99 years who match age within 5 years of cases and gender who do NOT have evidence of Paget's disease of bone as defined by:

  * No bone pain or bony deformity
  * Normal serum alkaline phosphatase

Exclusion Criteria:

* Osteosarcoma or other blastic bony metastases alone
* Fibrous dysplasia of bone
* Hyperostosis frontalis interna
* All men and women < 18 years or > 99 years
* Pregnancy (women) determined by self-report
* Current use of oral contraceptive tablets or Depo-Provera™ (women)
* Current use of hormone replacement therapy
* Creatinine clearance < 60 ml/min./1.73 m2 by Cockcroft-Gault based on most recent serum creatinine level (if greater than 1 year since last assessment, will be measured on collected blood sample to verify eligibility)
* Current smoking or tobacco use
* Alcohol use greater than 3 units daily
* Use of thiazolidinediones within the last year
* Use of medications known to impact bone and mineral metabolism, including use of a bisphosphonate in the last 11 months; ever use of teriparatide or denosumab; use of calcitonin, selective estrogen receptor modulators (SERMs), or estrogen within the past 6 months, prednisone > 5 mg for over 10 days in the last three months, anti-epileptic medications (e.g. phenytoin, carbamezapine, phenobarbitol, and primidone); current or use within the past year of aromatase inhibitors; leuprolide; histrelin
* History of a thyroid problem that is currently uncontrolled as defined by most recent thyroid stimulating hormone levels < 0.1 microIU/mL (if greater than 6 months since last assessment, will be measured on collected blood sample to verify eligibility)
* Other known metabolic or structural bone disease other than low bone density (e.g. hyperparathyroidism, multiple myeloma, sarcoid or other granulomatous disease, celiac disease, osteopetrosis, osteomalacia, osteitis fibrosa cystica)
* Other significant medical illness (heart disease, pulmonary disease, inflammatory bowel disease, malignancy other than ductal carcinoma in situ (DCIS) or non-melanoma skin cancer, rheumatologic conditions including rheumatoid arthritis, systemic lupus, renal disease requiring dialysis, etc.)
* Inability to understand and provide informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with active Paget's Disease of Bone but without other medical conditions or use of medications known to directly affect the bone. Healthy controls similar to age and gender will also be recruited.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-03 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Serum chemokine level | Day 1
  Compare the serum chemokine concentrations in research participants with Paget's disease of bone to research participants without Paget's disease of bone

SECONDARY OUTCOMES:
Correlation of chemokine level to Paget's Disease of Bone Pain | Day 1
  Correlate the serum chemokine concentration in research participants with Paget's disease of bone to burden of disease as assessed clinically by pain utilizing the Likert pain scale.
Correlation of chemokine level to alkaline phosphatase concentration | Day 1
  Correlate the serum chemokine concentration in research participants with Paget's disease of bone to burden of disease as assessed clinically by serum alkaline phosphatase concentration.
Correlation of chemokine level to proportion of affected skeleton | Day 1
  Correlate the serum chemokine concentration in research participants with Paget's disease to percent of skeleton affected as assessed radiographically by bone scan and x-ray.
Correlation of chemokine level to number of circulating stem cells | Day 1
  Correlate the serum chemokine concentration in research participants to number of circulating mesenchymal stem cell and epithelial progenitor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Crane, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided